CLINICAL TRIAL: NCT00267384
Title: N-acetylcysteine Protects From Aminoglycosides Induced Nephrotoxicity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Victor Novack, Head, Clinical research center, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sor407205ctil
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Drug Induced Nephrotoxicity
Keywords: Aminoglycosides
MeSH Terms: interventions — Acetylcysteine

INTERVENTIONS:
Drug: Oral N-Acetylcysteine

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial will be performed to assess the effect of N-acetylcysteine therapy on the incidence of nephrotoxicity among patients hospitalized with an infection and treated with aminoglycosides (AGs). Secondary goals of the study will be as follows: comparison of the mortality rates, and length of hospitalization among patients treated with N-acetylcysteine compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized with presumptive gram-negative infection, as assessed by the treating house staff and requiring gentamycin therapy according to an infectious disease specialist decision.
2. Aged between 18 and 90.
3. Recruitment time between starting gentamycin therapy and initiation of the study intervention will be less than 24 hours.
4. Signed informed consent.

Exclusion Criteria:

1. Any known allergy or intolerance to one of the medications in the AG group.
2. Any known allergy or intolerance to N-acetylcysteine.
3. Any immunosuppressive therapy excluding steroid therapy.
4. Pregnancy.
5. HIV infection.
6. Non-sepsis-related neutropenia.
7. An estimated creatinine clearance of less than 30 mL/min.
8. Acute renal failure defined as elevation in creatinine level of 0.5 mg/dL above the patient's baseline.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The decrease in glomerular filtration rate (GFR)

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Etzion, MD, Principal Investigator — Internal Medicine Division, Soroka University Medical Center; Victor Novack, MD, PhD, Principal Investigator — Internal Medicine Division, Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel